CLINICAL TRIAL: NCT04702360
Title: ELX/TEZ/IVA Expanded Access Program for Patients 6 Through 11 Years of Age With Cystic Fibrosis Who Have At Least One F508del Mutation
Brief Title: ELX/TEZ/IVA Expanded Access Program for Cystic Fibrosis (CF) Patients With at Least One F508del Mutation
Status: Approved for marketing | Type: Expanded Access
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX20-445-905
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination tablet for oral administration.
  Other Names: elexacaftor/tezacaftor/ivacaftor; VX-445/VX-661/VX-770
Drug: IVA — IVA monotablet for oral administration.
  Other Names: ivacaftor; VX-770

SUMMARY:
The purpose of this program is to provide elexacaftor/tezacaftor/ivacaftor (ELX/TEZ/IVA) to CF patients in critical need who are 6 to 11 years of age with at least one F508del mutation in response to unsolicited physician requests.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with confirmed diagnosis of CF who have an F/any genotype
* Prior treatment for at least 6 months with an approved alternative CFTR modulator (if the patient is eligible for such treatment)
* Patients with percent predicted forced expiratory volume in 1 second (ppFEV1) <40 for a minimum of 60 consecutive days before the date of completion of the request form

Key Exclusion Criteria:

* Patients with severe hepatic impairment

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 11 Years | Sex: All
Age Groups: Child